CLINICAL TRIAL: NCT05417360
Title: Effect of Pasteurized Akkermansia Muciniphilia on Maintenance of Body Weight After a Low Calorie Diet
Brief Title: Akkermansia and Weight Maintenance
Acronym: Amansia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NL80563.068.22
Record Dates: First submitted 2022-05-24; First posted 2022-06-14 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Obesity; Microtia; Metabolic Syndrome; Weight Loss
MeSH Terms: conditions — Obesity; Congenital Microtia; Metabolic Syndrome; Weight Loss

STUDY DESIGN:
Intervention Model Description: A double-blind, placebo-controlled randomised intervention study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized pasteurized A. muciniphila or placebo using variable block randomization with stratification for gender and age following the weight-loss period. The procedure will be done by an independent researcher using a validated variable block randomization model in the Castor database management system (DBMS). The same independent researcher will provide the participants with the supplements, and the product (pasteurized A. muciniphila or placebo). The supplement packages will not contain information about the content. Blinding will be maintained until the analysis has been completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Akkermansia muciniphila (A. muciniphila) (Experimental): After an 8-week low caloric diet (LCD, ~800kcal), participants who have successfully lost 8% of their body weight who are randomized to the intervention group, will receive pasteurized A. muciniphila.
  Interventions: Dietary Supplement: Akkermansia muciniphila
- Placebo (Placebo Comparator): After an 8-week low caloric diet (LCD, ~800kcal), participants who have successfully lost 8% of their body weight who are randomized to the control group, will receive a placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Akkermansia muciniphila — During the weight management period (weeks 8 to 32), the pasteurized A. muciniphila product will be orally consumed in water at least 15 min before breakfast for a period of 6 months (24 weeks) capsules. It appears as a white homogenous powder.
  .
  Arms: Akkermansia muciniphila (A. muciniphila)
Dietary Supplement: Placebo — During the weight management period (weeks 8 to 32), the placebo product will be orally consumed in water at least 15 min before breakfast for a period of 6 months (24 weeks). It appears as a white homogenous powder.
  Arms: Placebo

SUMMARY:
Obesity and related disorders such as type 2 diabetes are a worldwide diet-related problem. As such new treatment options are constantly being developed. Bacteria living in the gut seem to be a key player in the treatment of obesity and related metabolic diseases by influencing energy balance and the immune system. In terms of newly identified bacteria species, Akkermansia muciniphila (A. muciniphila) has been found to be related to obesity. Several animal studies have shown the beneficial impact of A. muciniphila on the treatment of body weight as well as insulin sensitivity.

The growth requirements of live A. muciniphila as well as its oxygen sensitivity rendered this bacterium unsuitable for human investigations or putative therapeutic opportunities. Therefore, pasteurization, a mild heating method, and its impact on diet-induced metabolic disorders in mice were investigated. Unexpectedly, this method of inactivation did not negate the effect of A. muciniphila, but improved its beneficial metabolic effects. Pilot studies have provided further evidence that pasteurization of A. muciniphila is safe for human use and has the potential to beneficially affect the control of body weight and glucose metabolism.

In this project, The investigators hypothesize that pasteurized A. muciniphila will be superior to placebo intervention in maintaining body weight after a phase of weight loss (low caloric diet) in adult participants with overweight or obesity.

DETAILED DESCRIPTION:
RATIONALE This study will examine the influence of specific beneficial gut bacteria in relation to weight maintenance. The worldwide prevalence of obesity, obesity-associated insulin resistance, and type 2 Diabetes Mellitus (T2DM) has grown dramatically over the last couple of decades; in every region of the world, obesity prevalence has more than tripled since 1975. Even though obesity treatment strategies, such as lifestyle interventions (focussed on diet and/or physical activity) and bariatric surgery have improved, there is extensive variability in responses. In the short term, reducing body weight is relatively easy, for most people. However, maintaining weight loss in the long term is a challenge. Hence, novel strategies to reduce these pandemics and support weight maintenance are strongly warranted.

The gut microbiome has emerged as an important regulator of host energy metabolism, thereby contributing to the etiology of obesity and obesity-related insulin resistance. However, scientific evidence is mainly derived from animal experiments and association studies, and support for causality in humans using mechanistic studies is limited. The influence of a newly identified bacterium, A. muciniphila. has been shown to be associated with a healthy intestine, and its abundance is inversely correlated to several disease states amongst others obesity and insulin resistance. However, the growth requirements of live A. muciniphila as well as its oxygen sensitivity(12) rendered this bacterium unsuitable for human investigations or putative therapeutic opportunities. Therefore, pasteurization, a mild heat inactivation method (30 min at 70 degrees Celsius), and its impact on diet-induced metabolic disorders in mice were investigated. Unexpectedly, this method of inactivation did not abolish the effect of A. muciniphila but even exacerbated its beneficial impacts. In mice, daily administration of pasteurized A. muciniphila alleviates diet-induced obesity. Moreover, a randomized, double-blind, placebo-controlled proof-of-concept study in overweight/obese insulin-resistant adults showed that the daily supplementation with pasteurized A. muciniphila for 12 weeks improved several metabolic parameters such as insulin sensitivity, insulinemia, plasma total cholesterol, as well as relevant blood markers for liver dysfunction and inflammation independently from any caloric restriction or modification of the physical activity. The investigators hypothesize that pasteurized A. muciniphila will be superior to placebo intervention in maintaining body weight after a low caloric diet in participants with overweight or obesity.

OBJECTIVES

1. To investigate the effects of pasteurized A. muciniphila on the maintenance of body weight after a phase of weight loss.
2. To investigate the effects of pasteurized A. muciniphila on body composition and body fat distribution, glucose homeostasis and insulin sensitivity, and metabolic health.
3. To investigate the effects of pasteurized A. muciniphila on the fecal bacterial composition and functionality, systemic inflammation, and gut barrier function and identify relevant biomarkers.

STUDY DESIGN The proposed study is a 32-week double-blind placebo-controlled randomized trial in 108 healthy overweight/ obese (BMI ≥ 28 kg/m2 < 40 kg/m2) Dutch adults, aged 20-70 years. All participants will follow a commercially-prepared low-calorie diet, with 15-20 energy % from fat, 35-40 energy % from protein, and 45-50 energy % from carbohydrates for a period of 8 weeks, to lose 8% of their body weight. In addition to these prepared meals, participants will be allowed limited consumption of specific low-calorie vegetables. Participants will be randomized to either the placebo or the intervention group following the weight-loss period. The weight loss phase will be followed by a 24-week supplementation placebo or active ingredient and a weight maintenance period. Prior to, as well as during both phases of the study participants will receive regular weigh-ins (weeks 0, 1, 4, 8, 16, 24, and 32) and counseling from a registered dietician. In addition to measuring changes in weight and physical measurements, participants will fill in questionnaires, and provide blood and fecal samples at weeks 0, 8, and 32.

QUALITY ASSURANCE Study activities will be carried out by qualified trained personnel, following standard operating procedures (SOP's). All research activities, including data entry and SOP compliance, will be monitored by an independent monitoring board, Clinical trial center Maastricht (CTCM). Data will be analyzed and handled according to the data management and statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 28 kg/m2 < 40 kg/m2
* Weight stable for at least 3 months (± 2 kg).

Exclusion Criteria:

* Type 2 diabetes mellitus (fasting plasma glucose ≥ 7.0 mmol/L)
* Gastroenterological diseases
* Surgery on the gastrointestinal tract (ex.Bariatric surgery)
* Cardiovascular diseases, cancer, liver or kidney malfunction, a disease with a life expectancy of < 5 years;
* Alcohol (>15 standard drinks per week) or drug abuse
* Excessive nicotine use is defined as >20 cigarettes per day;
* Use of prebiotics or probiotics 3 months prior to the start of the study;
* Intensive exercise training, > 3 hours a week;
* Use of any medication influencing glucose or fat metabolism (ex. lipid-lowering-drugs e.g. PPAR γ (peroxisome proliferator-activated receptors) or PPARα (fibrates) agonists), glucose-lowering agents (including all sulfonylureas, biguanides, α-glucosidase inhibitors, thiazolidinediones, repaglinide, nateglinide, and insulin), inflammation (e.g. anti-inflammatory or immunosuppressive drugs) and anti-oxidants);
* Regular use of laxatives
* Use of antibiotics in the last 3 months
* Vegan
* Lactose intolerance
* Pregnancy or lactation
* Concomitant participation in another study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Body weight | 6 months
  Changes in body weight following the initial weight loss period will be monitored over the weight maintenance period.

SECONDARY OUTCOMES:
Body composition | 8 months
  Changes in body composition following the initial weight-loss period as assessed by dual-energy X-ray absorptiometry (DEXA), and body mass index (BMI).
Body fat distribution | 8 months
  Changes in body fat distribution following the initial weight-loss period as assessed by the waist to hip ratio, as measured by waist and hip circumferences.
Glucose metabolism | 8 months
  Changes in glucose metabolism will be assessed by fasting glucose and hemoglobin A1C (HBA1c).
Insulin sensitivity | 8 months
  Changes in glucose and insulin responses to a 7 point oral glucose tolerance test.
Lipid profile | 8 months
  Changes in total cholesterol, triglycerides (TG), low-density lipoprotein) (LDL), high-density lipoprotein (HDL), and non - esterified fatty acids (NEFA) will be considered together to give an indication of the overall lipid profile as a result of the LCD and active intervention.
Adipose tissue activity | 8 months
  Changes in adipose tissue gene/protein expression will be assessed.
Gut barrier function | 8 months
  Gut barrier function will be assessed using serum/fecal zonulin, fecal calprotectin, serum LBP, and serum LPS. These measurements will be considered together to give an indication as to the function of the gut barrier, i.e. if it is normal, disrupted, or has improved as a result of the LCD and or active intervention.
Psychological well-being - mental health | 8 months
  Well-being, as it relates to feelings of depression and anxiety, will be measured using the Hospital Anxiety and Depression Scale (HADS) questionnaire.
Psychological well-being - sleep quality | 8 months
  Well-being, as it relates to sleep and sleep quality, will be assessed using the Pittsburgh Sleep Quality Index (PSQI)
Psychological well-being - stress | 8 months
  Well-being, as it relates to perceived stress, will be assessed using the 10-item Perceived Stress Scale (PSS).
Psychological well-being - General | 8 months
  general well-being will be assessed using the 36-Item Short-Form Health Survey (Rand - 36/ SF-36) .
Gastrointestinal symptoms - bowel movements | 8 months
  Gastrointestinal symptoms related to bowel movement frequency and consistency will be measured using the Bristol Stool Charts (BSC).
Gastrointestinal symptoms | 8 months
  Gastrointestinal symptoms will be measured using the Gastrointestinal Symptom Rating Scale questionnaire.
Heart rate | 8 months
  Changes in heart rate will be monitored over time
Blood pressure | 8 months
  Changes in blood pressure (systolic blood pressure (SBP), diastolic blood pressure (DBP)) will be measured over time.
Renal function | 8 months
  Changes in renal function, before during, and after the LCD and intervention will be monitored with blood creatinine, sodium, potassium, and chloride concentrations. These measurements will be considered together to determine if renal function is stable, has deteriorated, or improved.
Liver function | 8 months
  Changes in liver function will be monitored before during and after the LCD and active intervention using blood alanine aminotransferase (ALAT), aspartate transaminase (ASAT), alkaline phosphatase (ALP), gamma-glutamyltransferase (GGT), bilirubin, and, albumin. These measurements will be considered together to determine if liver function is stable, has deteriorated, or improved.
Inflammation | 8 months
  Inflammation will be monitored using C- reactive protein (CRP), lipopolysaccharide-binding protein (LBP), lipopolysaccharide (LPS), and serum zonulin.
Microbiota | 8 months
  Fecal samples to be used for analyzing microbiota composition will be collected and compared between groups.
Short chain fatty acid production | 8 months
  Circulating fatty acids will be measured as a measure of function of the microbiota

OTHER OUTCOMES:
Physical activity | 8 months
  Physical activity and sedentary behavior will be monitored using the Short QUestionnaire to ASsess Health-enhancing physical activity (SQUASH). The SQUASH measures the frequency, duration, and intensity of 4 different physical activities, namely physical activity to and from work, household activities, activities at work, and physical activities performed during free time. The higher the score, the more time is spent on physical activity.
Diet | 8 months
  Dietary intake will be monitored will be monitored using multiple 3 day weighed food diaries (food records)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Human Biology, Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
After completing the study, the generated data will be shared pseudo-anonymized (participant code, but no private data of the participants will be shared) with the subsiding party A-Mansia Biotech. There are no restrictions with respect to the publication of the data. Both positive and negative results of the studies will be made public, preferably in peer-reviewed international scientific journals, according to the Central Committee on Research involving Human Subjects (CCMO) statement of publication policy. The authorship of the article shall be determined with consideration based on the contribution to the set-up and execution of the study and active participation in publication. Further, this study will be registered in a public trial registry before the first volunteer will be recruited.